CLINICAL TRIAL: NCT01553162
Title: B-precursor Acute Lymphoblastic Leukemia (ALL): Studying the Mechanisms Behind Dexamethasone and Prednisone Sensitivity in High-Risk Patients
Brief Title: Studying Dexamethasone and Prednisone Sensitivity in Samples From Younger Patients With High-Risk B-Cell Precursor Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AALL12B4; COG-AALL12B4 (Other: Children's Oncology Group); CDR0000728515 (Other: clinicaltrials.gov); AALL12B4 (Other: COG); NCI-2012-00704 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-03-10; First posted 2012-03-14 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: B-cell childhood acute lymphoblastic leukemia; untreated childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia | interventions — Gene Expression Profiling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: RNA analysis
Genetic: gene expression analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood, tissue, or bone marrow from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research trial is studying dexamethasone and prednisone sensitivity in samples from younger patients with high-risk B-cell precursor acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify differences in the effect of dexamethasone (Dex) and prednisone (Pred) on glucocorticoid receptor (GR) occupancy and gene expression in high-risk (HR) B-cell precursor (BCP)-acute lymphoblastic leukemia (ALL) samples from patients aged 1-9.
* Identify differences in gene expression and GR occupancy of response elements in HR BCP-ALL patients > 10 years old in response to both Dex and Pred.

OUTLINE: Archived samples are analyzed for gene expression analysis and genomic location of glucocorticoid receptor by ChIP sequencing (ChiPseq) and RNA sequencing. Data of gene expression and ChiPseq data sets are compared by luciferase reporter assay.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients diagnosed with high-risk B-cell precursor acute lymphoblastic leukemia
* Samples from patients treated and not treated with Dex and Pred

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients diagnosed with high-risk B-cell precursor acute lymphoblastic leukemia
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-04; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Differentially expressed genes from both HR BCP-ALL patients aged 1-9 and patients over 10 years old
Genes that are required for efficient apoptosis

CONTACTS AND LOCATIONS:
Overall Officials: Miles A. Pufall, PhD, Principal Investigator — University of Iowa